CLINICAL TRIAL: NCT07250737
Title: Managed Access to Investigational Use of AOC 1044 in Participants With DMD Mutations Amenable to Exon 44 Skipping
Brief Title: Managed Access Program for Del-zota in Participants With DMD Mutations Amenable to Exon 44 Skipping
Status: Available | Type: Expanded Access
Sponsor: Avidity Biosciences, Inc. (Industry)
Collaborators: Clinigen Healthcare Limited (Unknown)
Responsible Party: Sponsor
Other Study IDs: AOC 1044-MAP
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Muscular Disorders, Atrophic; Muscular Diseases; Musculoskeletal Diseases; Neuromuscular Diseases; Nervous System Diseases; Genetic Diseases, Inborn; Genetic Diseases, X-Linked; Muscular Dystrophies; Muscular Dystrophy, Duchenne
Keywords: Avidity; Avidity Biosciences; AOC 1044; AOC 1044-CS1; AOC 1044-CS2; EXPLORE44; EXPLORE44-OLE; Del-zota; delpacibart zotadirsen; DMD; exon skipping therapy; dystrophin; managed access; expanded access; pre-approval access; compassionate use; MAP; EAP
MeSH Terms: conditions — Muscular Disorders, Atrophic; Muscular Diseases; Musculoskeletal Diseases; Neuromuscular Diseases; Nervous System Diseases; Genetic Diseases, Inborn; Genetic Diseases, X-Linked; Muscular Dystrophies; Muscular Dystrophy, Duchenne

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: delpacibart zotadirsen — Del-zota is administered as an IV infusion every 6 weeks. Doses are administered based on body weight.
  Other Names: Del-zota; AOC 1044

SUMMARY:
The purpose of this Managed Access Program is to allow access to delpacibart zotadirsen (AOC 1044) for eligible patients diagnosed with DMD mutations amenable to exon 44 skipping. The patient's Administering Physician should follow the suggested treatment guidelines and comply with all local health authority regulations.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be permanently residing in the US and have a US primary health care provider.
* Documented dystrophin gene mutation that is amenable to exon 44 skipping.
* Age 6 or older at the time of consent.
* Participants must be willing to use effective contraception methods (e.g., abstinence, condom with or without spermicide) if engaged in sexual relations.
* The participant must be able to provide written and dated informed consent and/or assent, where applicable, prior to participating in any program procedures. The informed consent and assent processes will be conducted in accordance with local IRB guidelines and applicable local/national laws.
* Participants who have been previously treated with a gene therapy for DMD can be eligible if in the opinion of the administering physician, have had an unsatisfactory treatment response AND the treatment with gene therapy and associated immunosuppressive regimen was received more than 12 months before informed consent signing.

Exclusion Criteria:

* Participation in a clinical study in which the participant received an investigational drug within 30 days, 5 half-lives, or twice the duration of the biological effect of the investigational drug, whichever is longest, prior to informed consent.
* Participants with any of the following, despite being on optimal medical management: serious respiratory dysfunction (history of continuous invasive respiratory support), or significant cardiac dysfunction (LVEF < 40%), or nearing end of life.
* eGFR <75 mL/min/1.73 m2 as calculated by CKiD formula (see https://kidney.wiki/gfr-calculator).
* Participants who discontinued early from the treatment period of the EXPLORE44 (CS1) or EXPLORE44-OLE (CS2) trials.

Min Age: 6 Years | Sex: Male
Age Groups: Child, Adult, Older Adult
Gender Based: Yes